CLINICAL TRIAL: NCT07217353
Title: The Use of a Novel Vaginal Speculum for Endometrial Biopsies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rocky Vista University, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-158
Record Dates: First submitted 2025-10-03; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Endometrial Cancer
Keywords: Endometrial biopsies; Endometrial Cancer; Vaginal Speculum
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Endometrial biopsies with a new vaginal speculum (Experimental): The use of a novel, FDA-cleared vaginal speculum for endometrial biopsies
  Interventions: Device: Bouquet Speculum

INTERVENTIONS:
Device: Bouquet Speculum — Novel Bouquet Speculum used for endometrial biopsies

SUMMARY:
The objective of this clinical trial is to determine if a newly-designed and FDA-cleared vaginal speculum (the Bouquet Speculum) will provide better visualization of the cervical os, be easier and more efficient to use, provide more consistent outcomes and decrease the discomfort associated with endometrial biopsy procedures.

DETAILED DESCRIPTION:
To answer the question, "How does the Bouquet speculum compare to a two-bladed speculum in terms of patient comfort, provider visualization, ease of use, and accuracy for obtaining samples for in-office endometrial biopsies for patients with endometrial cancer requiring follow up procedures?" the investigators will have an observational study of 100 women aged 18-90 years old that have previously had an endometrial biopsy with the use of a two-bladed speculum. Providers (physicians, physician's assistants, and nurse practitioners) at Minnesota Oncology Clinics will be educated on how to use the Bouquet speculum via a Zoom training session, a video presentation, and step-by-step instructional page that has been used in previous studies on the product. The providers will use the Bouquet speculum for endometrial biopsies on patients that consent to the study that come into the clinic for the procedure. The providers will do the procedures in the same way as they usually do but will use the Bouquet speculum instead of a two-bladed speculum.

To analyze the question, this research will measure the variables of patient comfort level, and provider ease-of-use with the Bouquet speculum, the extent of visualization of the cervix, and accuracy of sampling of the endometrium lining (the necessary result of an endometrial biopsy). The variables of patient weight and parity will be included in the patient survey to determine if they have an effect on the outcomes of visualization, ease-of-use, accuracy of sampling, and patient comfort level.These measurements will be recorded via a survey for the patient and provider following the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Biological women with a uterus, age 18-90
* Previous endometrial biopsy procedure performed at the Minnesota Oncology Clinic

Exclusion Criteria:

* Pregnant women, active pelvic infection, or uncontrolled bleeding dyscrasias as determined by the provider at Minnesota Oncology Clinics
* Biological women without a uterus who are less than 18 years old or greater than 90 years old, or who have not had a previous endometrial biopsy at the Minnesota Oncology Clinic.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological females with an intact uterus who may identify as male
Enrollment: 100 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Provider visualization of the cervix, ease of use, and accuracy of a new vaginal speculum being used for endometrial biopsies | Through study completion, an average of 1 year
  A simple survey is filled out by the provider regarding whether the visualization of the cervix was better, the same, or worse with the new vaginal speculum. Similarly, the provider will be asked on the survey about the ease of use (easier, same more difficult). The last criteria will be de-identified data from the cohort to see if an adequate sample was obtained of the endometrium.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Dement, MA, Study Director — Rocky Vista University

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: October 2025-October 2026
Access Criteria: Statistical analysis will be performed at RVU through Dr. Mark Payton. Any data that is shared will require a data sharing agreement.
URL: http://www.rvu.edu

REFERENCES:
- [Result] Luzarraga Aznar A, Canton R, Loren G, Carvajal J, de la Calle I, Masferrer-Ferragutcasas C, Serra F, Bebia V, Bonaldo G, Angeles MA, Cabrera S, Palomar N, Vilarmau C, Marti M, Rigau M, Colas E, Gil-Moreno A. Current challenges and emerging tools in endometrial cancer diagnosis. Int J Gynecol Cancer. 2025 Apr;35(4):100056. doi: 10.1016/j.ijgc.2024.100056. Epub 2024 Dec 18. PMID 40011116
- [Result] Amant F, Moerman P, Neven P, Timmerman D, Van Limbergen E, Vergote I. Endometrial cancer. Lancet. 2005 Aug 6-12;366(9484):491-505. doi: 10.1016/S0140-6736(05)67063-8. PMID 16084259
- [Result] Khan S, Waters-Kellar L, Barsh E, Shannon A, Clark S, Ryznar RJ, Trawick A, Payton M, Bouquet J. A Survey of Physicians and Patients in Pakistan Assessing the Improvement of Visualization of the Cervix, Ease of Use, and Patient Comfort Using a Newly Designed Vaginal Speculum: A Pilot Study. Med Devices (Auckl). 2025 Jun 11;18:309-317. doi: 10.2147/MDER.S509134. eCollection 2025. PMID 40599808
- [Result] Bouquet JM, Morris E, Zapata I. A novel and cost-effective model to screen and treat cervical cancer and precancers at the point of care. Front Public Health. 2025 Apr 16;13:1527172. doi: 10.3389/fpubh.2025.1527172. eCollection 2025. PMID 40308928
- [Result] Bouquet JM, Naji R, Armas CA, Roldan V, Selkhi S, Bentley CZ, Zapata I, Fisher J. An Innovative Design for the Vaginal Speculum. Med Devices (Auckl). 2023 Sep 25;16:211-218. doi: 10.2147/MDER.S415558. eCollection 2023. PMID 37790696
- Available data/document: Study Protocol: IRB 2025-158 — https://www.axiommentor.com/pages/irb/sectionsOfProtocol.cfm?id=977&b=MP